CLINICAL TRIAL: NCT06238713
Title: Extraperitoneal SINgle-port rObotic-assisted Radical Prostatectomy (RARP) Versus Transperitoneal Multi-port RARP in the Treatment Of Prostate Cancer (SINO-TOP)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); ShuGuang Hospital (Other); Eastern Hepatobiliary Surgery Hospital (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); Sir Run Run Shaw Hospital (Other); Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Ren Shancheng, Professor，Chief of Urology, Shanghai Changzheng Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SINO-TOP-23
Record Dates: First submitted 2024-01-15; First posted 2024-02-02 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Prostate Adenocarcinoma; Localized Prostate Carcinoma
Keywords: Prostate Cancer; Robotic-assisted Radical Prostatectomy; da Vinci surgical robot; Potency; Non-inferiority; RCT; Continence
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single-port extraperitoneal RARP (Experimental): Single-port extraperitoneal robotic-assisted radical prostatectomy with Vattikuti Institute Prostatectomy (VIP) techniques
  Interventions: Procedure: Single-port extraperitoneal robotic-assisted radical prostatectomy with Vattikuti Institute Prostatectomy（VIP） techniques
- Multi-port transperitoneal RARP (Active Comparator): Multi-port transperitoneal RARP with bilateral intrafascial nerve-sparing techniques
  Interventions: Procedure: Multi-port transperitoneal robotic-assisted radical prostatectomy with bilateral intrafascial nerve-sparing techniques

INTERVENTIONS:
Procedure: Single-port extraperitoneal robotic-assisted radical prostatectomy with Vattikuti Institute Prostatectomy（VIP） techniques — Patients with localized prostate cancer are randomized into this group in a 1:1 ratio and receive single-port extraperitoneal robotic-assisted radical prostatectomy with Vattikuti Institute Prostatectomy（VIP） techniques. The investigators will monitor patients for perioperative data recording, treatment and 1-year follow-up.
  Arms: Single-port extraperitoneal RARP
Procedure: Multi-port transperitoneal robotic-assisted radical prostatectomy with bilateral intrafascial nerve-sparing techniques — Patients with localized prostate cancer are randomized into this group in a 1:1 ratio and receive multi-port transperitoneal robotic-assisted radical prostatectomy with bilateral intrafascial nerve-sparing techniques. The investigators will monitor patients for perioperative data recording, treatment and 1-year follow-up.
  Arms: Multi-port transperitoneal RARP

SUMMARY:
This study is a two-arm, multicenter, randomized controlled clinical trial on whether single-port extraperitoneal VIP RARP is non-inferior to multi-port transperitoneal RARP in terms of functional recovery rate and other key metrics.

DETAILED DESCRIPTION:
Multicenter enrollment of 480 patients with localized prostate cancer meeting enrollment criteria are randomized to undergo either single-port robotic extraperitoneal VIP radical prostatectomy or multi-port robotic transperitoneal bilateral intrafascial radical prostatectomy for perioperative data recording, treatment, and monitoring with 1 year follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Men aged 18 years ≤ age ≤ 75 years;
2. Prostate biopsy within 6 months with diagnosis of organ-localized prostate cancer with preoperative staging of T1c to T2b,N0M0;.
3. Gleason Score<8.
4. PSA<20ng/ml.
5. Pathologic diagnosis of prostate follicular adenocarcinoma or prostate ductal adenocarcinoma;
6. The patient has healthy sexual function before surgery and intention for sexual activities after surgery;
7. Physiological condition acceptable for laparoscopic surgery;
8. Willing to cooperate and complete the study follow-up and related examinations;
9. The subject or his agent voluntarily participates in this trial and signs the written informed consent;
10. The questionnaire can be completed in Chinese.
11. The patient has been informed of the trial;

Exclusion Criteria:

1. High-risk and non-organ localized prostate cancer (clinical stage ≥ T2c, GS ≥ 8, PSA > 20ng/ml);
2. Special type of prostate cancer， such as neuroendocrine etc.;
3. History of previous abdominal surgery and radiotherapy which may affect abdominal incision and Port placement;
4. Recent surgery of rectum, perianal abscess or around fistula and perineal area;
5. Patients who have undergone previous electro-prostatectomy/enucleation of the prostate;
6. Non-recurrent patients with less than 12 months of follow-up;
7. ECOG>1.
8. Combination of other systemic tumors;
9. had received any type of preoperative antitumor therapy;
10. Suffering from poor general condition with the presence of one of the following conditions: including severe mental disorders, cardiovascular disease, active infections, bone marrow transplantation within 3 months, or significant abnormalities in organ function;
11. Participation in other clinical studies or previous treatment with any gene therapy product within the last 3 months;
12. Other conditions that the researchers believe may affect the experimental results or are unethical;

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Potency recovery rate | 3 months after surgery
  Potency recovery rate 3 months postoperatively, based on the patient's description of whether the erection is firm enough for sexual activity or intercourse.

SECONDARY OUTCOMES:
Continence recovery rate | Up to 1 year, at a frequency of 1, 3, 6, and 12 months postoperatively
  The rate of recovery of continence postoperatively, measured in the number of pads used per day.
PSA | Up to 1 year, at a frequency of 1, 3, 6, and 12 months postoperatively
  PSA status postoperatively，measured in ng/mL
Potency recovery rate | Up to 1 year, at a frequency of 1, 6, and 12 months postoperatively
  Potency recovery rate will be assessed by patient's self-reported erectile firmness for sexual activity or intercourse, International Index of Erectile Dysfunction(IIEF-5) score（from 0-25 score, a higher score means a worse outcome）, and phosphodiesterase5 (PDE-5）inhibitor intake frequency according to patients' despciption (a higher intake means a worse outcome）.
Clavien-Dindo complication score | Every day during period of hospitalization (up to 7 days)
  Clavien-Dindo complication score measured in the following grades（a higher grade means a worse outcome） ： First grade：complications that do not require medication, surgery or endoscopic treatment.
  Second grade： complications require to be treated with drugs, including blood transfusion and parenteral nutrition.
  Third grade： complications that require surgery, endoscopy, or radiation therapy.
  Fourth grade: the emergence of life-threatening complications, including cerebral hemorrhage, etc., which is also divided into 4a and 4b, 4a is single-organ dysfunction, 4b is mainly multi-organ dysfunction and injury.
  Fifth grade: death.
Operative time | During operation（on an average of 90-120minutes ）
  Time elapsed from skin incision to placement of the final skin suture, measured in minutes
Estimated blood loss | During operation（on an average of 90-120minutes ）
  Estimated blood loss, measured in volume (mL)
Number of additional ports | During operation（on an average of 90-120minutes ）
  Number of additional ports needed in surgery
Period of hospitalization | During period of hospitalization (up to 7 days)
  Hospital stay, counted in days from the first day of hospitalization to discharge
Period of hospitalization post surgery | Post surgery, during period of hospitalization (up to 7 days)
  Hospital stay, counted in days from the time of transfer to the post anesthesia care unit (PACU) to discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Changzheng hospital, Shanghai, Shanghai Municipality, China